CLINICAL TRIAL: NCT05947279
Title: Examining Lateralized Aspects of Motor Control Using Non-invasive Neural Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HM20025761
Record Dates: First submitted 2023-06-30; First posted 2023-07-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Motor Adaptation and Generalization; Posterior Parietal Cortex; Cerebellum

STUDY DESIGN:
Intervention Model Description: The study will have three groups: (15 people per group) 1) posterior parietal cortex group, which will receive the stimulation to their left posterior parietal cortex, 2) cerebellum group, which will receive stimulation to their right cerebellum, and 3) sham group, which will have the electrode cap placed on their head but receive no stimulation. By comparing motor adaptation reaching performance between these three groups, the investigators can examine how stimulation to each specific area of the brain modulates different aspects of motor adaptation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Posterior parietal cortex group (Experimental): Posterior parietal cortex group, which will receive the stimulation to their left posterior parietal cortex
  Interventions: Behavioral: Comparing motor adaptation reaching performance
- Cerebellum group (Experimental): Cerebellum group, which will receive stimulation to their right cerebellum,
  Interventions: Behavioral: Comparing motor adaptation reaching performance
- Sham group (Sham Comparator): Sham group, which will have the electrode cap placed on their head but receive no stimulation
  Interventions: Behavioral: Comparing motor adaptation reaching performance

INTERVENTIONS:
Behavioral: Comparing motor adaptation reaching performance — By comparing motor adaptation reaching performance between these three groups, the investigators can examine how stimulation to each specific area of the brain modulates different aspects of motor adaptation

SUMMARY:
Motor adaptation and generalization are believed to occur via the integration of various forms of sensory feedback for a congruent representation of the body's position in space along with estimation of inertial properties of the limb segments for accurate specification of movement. Thus, motor adaptation is often studied within curated environments incorporating a "mis-match" between different sensory systems (i.e. a visual field shift via prism googles or a visuomotor rotation via virtual reality environment) and observing how motor plans change based on this mis-match. However, these adaptations are environment-specific and show little generalization outside of their restricted experimental setup. There remains a need for motor adaptation research that demonstrates motor learning that generalizes to other environments and movement types. This work could then inform physical and occupational therapy neurorehabilitation interventions targeted at addressing motor deficits.

DETAILED DESCRIPTION:
Voluntary movement and sensory perception are fundamental aspects of the human experience. Senses such as visual and proprioceptive feedback inform movement by continuously providing the central nervous system with information on limb location, movement error, and task performance. However, the specific mechanisms behind how different forms of sensory information are used to adapt and generalize movement remain poorly understood.

Motor adaptation, or the modification of movement based on error feedback (Martin et al., 1996), is often elicited during rehabilitation but must be generalized to functional performance, such as activities of daily living, in order to successfully rehabilitate motor deficits following stroke. Motor adaptation and generalization are believed to occur via the integration of various forms of sensory feedback for a congruent representation of the body's position in space along with estimation of inertial properties of the limb segments for accurate specification of movement. Thus, motor adaptation is often studied within curated environments incorporating a "mis-match" between different sensory systems (i.e. a visual field shift via prism googles or a visuomotor rotation via virtual reality environment) and observing how motor plans change based on this mis-match. However, these adaptations are environment-specific and show little generalization outside of their restricted experimental setup. There remains a need for motor adaptation research that demonstrates motor learning that generalizes to other environments and movement types. This work could then inform physical and occupational therapy neurorehabilitation interventions targeted at addressing motor deficits.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed as determined by the short-form Edinburgh Handedness Inventory
* Between the ages of 18 and 40

Exclusion Criteria:

* Mixed- or left-handed as determined by the short-form Edinburgh Handedness Inventory
* Self-reported history of any of the following:

Seizure and/or diagnosis of epilepsy Fainting spells Concussion with loss of consciousness Ringing in the ears (tinnitus) Cochlear implants Migraines Diagnosed psychological or neurological condition Metal in the scalp

* Any previous adverse reaction to a brain stimulation technique
* Any previous adverse reaction to 3D virtual reality environments (i.e. 'cybersickness')
* Possibility of being currently pregnant (for females only)
* Current open head wound or skin condition of the scalp
* Current implanted device(s) (i.e. cardiac pacemaker)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Initial direction error, or difference between participant's fingertip direction | Completion of the study visit, approx 20 minutes
  Initial direction error, or difference between participant's fingertip direction at the timepoint of peak velocity relative to a linear path to the target. As for time frame, this is a single-visit study. Initial direction error will be compared during baseline reaching and following 20 minutes of non-invasive neural stimulation.
Initial direction error variance | Completion of the study visit, approx 20 minutes
  Initial direction error variance across multiple trials.

SECONDARY OUTCOMES:
Final position error | Completion of the study visit, approx 20 min
  Secondary outcome: final position error, or distance from participant's fingertip position at the conclusion of the reach to the center of the target. Similar to above, this measure will be compared during baseline and following 20 minutes of stimulation.
Final position error variance across multiple trials. | Completion of the study visit, approx 20 min
  Final position error variance across multiple trials.
Deviation from linearity | Completion of the study visit, approx 20 min
  Deviation from linearity, or a ratio of minimum and maximum displacement across the parallel and perpendicular planes of the reaching movement.
Peak tangential velocity | Completion of the study visit, approx 20 min
  Peak tangential velocity, or highest tangential velocity reached during reach.

CONTACTS AND LOCATIONS:
Locations (1):
- Virginia Commonwealth University Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No